CLINICAL TRIAL: NCT06711705
Title: Phase II MRD-Adapted Study of Elranatamab in Relapsed/Refractory
Brief Title: Elranatamab in Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ah-Reum "Autumn" Jeong, Assistant Clinical Professor, Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810312
Record Dates: First submitted 2024-11-12; First posted 2024-12-02 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elranatamab
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Phase II, single arm, open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elranatamab (Experimental): Treatment with elranatamab
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Subcutaneous injection of elranatamab. If patient achieves MRD negative remission, patient would enter treatment-free observation period with MRD monitoring.
  Other Names: Elrexfio

SUMMARY:
This study evaluates the efficacy of elranatamab alone in patients with relapsed and/or refractory Multiple myeloma who has previously received 1 to 3 combinations of treatment.

DETAILED DESCRIPTION:
Phase II study of elranatamab in patients with relapsed/refractory multiple myeloma who has received 1 to 3 prior lines of therapy. Patients may enter treatment-free observation period if they have a sustained MRD negative response for greater than 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Prior diagnosis of relapsed/refractory MM and have received 1 to 3 prior lines of therapy as defined by the IMWG criteria (Rajkumar et al., 2014) including anti-CD38 monoclonal antibody, proteosome inhibitor (PI), and immunomodulatory drug (IMiD), and BCMA-directed chimeric antigen receptor T-cell (CAR T-cell) therapy

   1. Refractory is defined as having disease progression while on therapy or within 60 days of last dose in any line, regardless of response.
   2. If participant has not received BCMA-directed CAR T-cell therapy, must be ineligible for CAR T-cell therapy or deferred such treatment by participant
4. Aged greater or equal to 18 years
5. Measurable disease as defined by any of the following:

   1. Serum M-protein level ≥ 0.5 g/dL by serum protein electrophoresis (SPEP), or
   2. Urine M-protein ≥ 200mg/24 hours by urine protein electrophoresis (UPEP), or
   3. Involved serum free light chain ≥ 10 mg/dL (≥100mg/L) AND an abnormal serum free light chain ratio in patients without measurable disease in the serum or urine
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
7. Adequate hematological function defined as

   1. Absolute neutrophil count (ANC) ≥1,000/mm3 (G-CSF not permitted for at least 1 week prior to the first dose of elranatamab)
   2. Hemoglobin ≥8.0 g/dL (transfusion support is permitted if completed at least 1 week prior to planned start of dosing)
   3. Platelet count ≥75,000/mm3 or ≥50,000/mm3 if >50% involvement with plasma cells in the screening bone marrow (transfusion support is permitted if completed at least 1 week prior to planned start of dosing)
8. Adequate renal function with estimated creatinine clearance (CrCl) ≥30 mL/min as calculated using Cockcroft-Gault equation.
9. Adequate liver function defined as

   1. Aspartate and alanine aminotransferase (AST and ALT) ≤2.5 x upper limit of normal (ULN); ≤5.0 x ULN if there is liver involvement by the tumor.
   2. Alkaline phosphatase ≤2.5 x ULN (≤5 x ULN in case of bone metastasis).
   3. Total bilirubin ≤2.0 mg/dL, except in patients with Gilbert Syndrome who must have a total bilirubin less than 3.0 mg/dL.
10. Able to receive outpatient treatment of elranatamab by meeting the following criteria:

    1. Lives within 30minutes from the site of medication administration
    2. Reliable caregiver present, who is able to watch participant continuously for at least until 48 hours after administration of first full treatment dose
    3. No history of grade 3-4 CRS or grade 3-4 ICANS from other immune effector cell or bispecific antibody therapies
11. Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1
12. Serum pregnancy test (for females of childbearing potential) negative at screening.

    a. Female patients of non-childbearing potential must meet at least 1 of the following criteria: i. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state.

    ii. Have undergone a documented hysterectomy and/or bilateral oophorectomy. iii. Have medically confirmed ovarian failure. b. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.
13. Agreement to adhere to Lifestyle Considerations (see section 5.3 and Appendix 2) throughout study duration

Exclusion Criteria:

1. Subjects with smoldering multiple myeloma, IgM multiple myeloma, Waldenstrom's macroglobulinemia, amyloidosis, POEMS syndrome, and primary and secondary plasma cell leukemia, defined as circulating plasma cells ≥ 5%
2. Extramedullary relapse who does not meet criteria for measurable disease as above
3. Active malignancy other than Multiple Myeloma requiring treatment in the past 3 years, with the exception of successfully treated non-metastatic squamous or basal skin carcinoma
4. Known CNS involvement by multiple myeloma
5. Active, uncontrolled autoimmune disorders
6. Active uncontrolled infection. Active infections must be resolved and/or controlled at least 14 days prior to enrollment.
7. Radiation therapy within 2 weeks prior to study entry (bone lesions requiring radiation may be treated with limited [ie, ≤25% of bone marrow in field] radiation therapy during this period).
8. Last systemic treatment within 2 weeks or 5 half lives, whichever is shorter. Subjects can receive a maximum of 160mg of dexamethasone or equivalent during screening, but at least 7 days prior to start of therapy.
9. Last radiation treatment to multiple sites within 2 weeks and single site within 1 week
10. History of autologous stem cell transplant within 100 days prior to study enrollment.
11. History of allogeneic transplant within 1 year prior to study enrollment or active graft versus host disease.
12. On immunosuppressive therapy for concurrent comorbid conditions
13. Other major uncontrolled medical comorbidities that may put patients at risk of serious adverse event with treatment with study medication.
14. Clinically significant, uncontrolled cardiac disease
15. Grade ≥2 peripheral sensory or motor neuropathy
16. History of Guillan-Barre syndrome
17. Other surgical (including major surgery within 14 days prior to enrollment) or psychiatric conditions including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
18. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
19. Pregnancy or lactation
20. Known or suspected hypersensitivity to the study intervention or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate as best response | 1 year of starting treatment
  MRD negativity rate as best response

SECONDARY OUTCOMES:
Sustained MRD negativity rate at 10^-5 | Through study completion, up to 5 years
  Sustained MRD negativity rate at 10^-5
Overall response rate | Within 1 year of treatment
  Overall response rate
Complete response rate | Within 1 year of treatment
  Complete response rate
Progression free survival | Through study completion, up to 5 years
  Progression free survival
Duration of response | Through study completion, up to 5 years
  Duration of response
Safety (cytokine release syndrome, neurotoxicity, treatment-related adverse events) | Through study completion, on average 4 weeks (cytokine release syndrome, neurotoxicity); Through study completion, up to 5 years (treatment-related adverse events as assessed by CTCAE v5.0 )
  Number of participants with cytokine release syndrome, neurotoxicity, treatment-related adverse events as assessed by CTCAE v5.0
Quality of life (questionnaire and by EORTC QLQ-MY20 questionnaire) | Through study completion, up to 5 years
  Quality of life assessed by cancer therapy satisfaction questionnaire and by EORTC QLQ-MY20 questionnaire

OTHER OUTCOMES:
Soluble BCMA, T-cell immune phenotype | 1 year
  Soluble BCMA, T-cell immune phenotype
Overall MRD negativity rate at 10^-6 | 1 year
  Overall MRD negativity rate at 10^-6

CONTACTS AND LOCATIONS:
Overall Officials: Ah-Reum Jeong, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States